CLINICAL TRIAL: NCT01752998
Title: Treating Chronic Pain in Buprenorphine Patients in Primary Care Settings
Acronym: BupPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA032800; 1205-002 (Other: Butler Hospital)
Record Dates: First submitted 2012-12-17; First posted 2012-12-19 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Pain; Depression; Substance Use
Keywords: pain; depression; substance use
MeSH Terms: conditions — Pain; Depression; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TOPPS Intervention (Active Comparator): Individuals randomized into this arm will receive 7 individual sessions of the Treating Opioid Patients' Pain and Sadness (TOPPS) intervention, designed to reduce symptoms of pain and depression.
  Interventions: Behavioral: Treating Opioid Patients' Pain and Sadness (TOPPS)
- Health Education (Placebo Comparator): Individuals randomized into this arm will receive 7 individual sessions on general health education.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Treating Opioid Patients' Pain and Sadness (TOPPS)
  Arms: TOPPS Intervention
Behavioral: Health Education
  Arms: Health Education

SUMMARY:
Individuals will be recruited by posted advertisements in the waiting rooms of the PCP offices and by physician referral. After an initial phone screen, research staff will meet with interested individuals in their PCP offices for informed consent, baseline interview and randomization. Participants will be randomized into a Health Education study arm, and receive 7 individual sessions on general health education, or an Intervention study arm, and receive 7 individual sessions of the Treating Opioid Patients' Pain and Sadness (TOPPS) intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Pain, defined as pain duration for at least six months with a mean score of 5 or higher on the BPI Pain Interference Scale;
* Pain severity of 40 or higher on a Visual Analog Scale (0-100) indicating "worst pain in the last week";
* Previous attempt at initial steps of PCP guideline pain care: must have had at least one trial of recommended medication (i.e. acetaminophen, NSAIDS, skeletal muscle relaxants) judged through interviews with patients and PCPs;
* QIDS score of ≥ 10 (depression severity)
* If using an antidepressant, the dose must be stable for the previous 2 months;
* Age 18 or older
* Has received buprenorphine/naloxone (Suboxone)for at least the last 3 months;
* Plan to continue buprenorphine/naloxone (Suboxone)for at least 3 months.

Exclusion Criteria:

* Lifetime DSM-IV diagnosis of bipolar disorder, schizophrenia, or other chronic psychotic condition;
* Current DSM-IV diagnosis of substance dependence for sedative/hypnotic drugs, alcohol, stimulants, or cocaine;
* Suicidal ideation or behavior requiring immediate attention;
* In psychotherapy or in a multidisciplinary pain management program at baseline;
* Anticipate having surgery in the next 6 months;
* Pain thought to be due to cancer, infection, inflammatory arthritis, or associated with severe or progressive neurological deficits;
* SSDI or SSI claim pending;
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Pain | 4 months
  Pain, as measured by self-report

SECONDARY OUTCOMES:
Depression | 4 months
  Depression, as measured by self-report and clinician-administered assessments
Substance Use | 4 months
  Illicit substance use, as measured by self-report and urine toxicology

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States